CLINICAL TRIAL: NCT05279183
Title: Assessment of Reward Responses to Erythritol Using Flavor Preference Learning and Its Effects on Gastrointestinal Hormones, Glycemic Control, Appetite-related Sensations and Emotional State
Brief Title: Assessment of Reward Responses to Erythritol Using Flavor Preference Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PolyReward
Record Dates: First submitted 2022-02-14; First posted 2022-03-15 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Reward Responses; Gastrointestinal Hormones; Glycemic Control; Appetite; Satiation; Emotional State
MeSH Terms: interventions — Erythritol; Sucrose; trichlorosucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Erythritol (Active Comparator): 20 volunteers receive erythritol dissolved in 300 mL tap water as oral preloads (3 times 100mL). The dosage will be calculated based on the participants ratings of the sweetness intensity (matched sweetness to 10 % sucrose).
  Interventions: Dietary Supplement: Erythritol
- Sucrose (Active Comparator): 20 volunteers receive 30g sucrose dissolved in 300 mL tap water as oral preloads (3 times 100mL).
  Interventions: Dietary Supplement: Sucrose
- Sucralose (Active Comparator): 20 volunteers receive sucralose dissolved in 300 mL tap water as oral preloads (3 times 100mL). The dosage will be calculated based on the participants ratings of the sweetness intensity (matched sweetness to 10 % sucrose).
  Interventions: Dietary Supplement: Sucralose

INTERVENTIONS:
Dietary Supplement: Erythritol — Subject specific dose of erythritol dissolved in 300 mL tap water.
  Other Names: E968-Erythritol
  Arms: Erythritol
Dietary Supplement: Sucrose — 30 g sucrose dissolved in 300 mL tap water.
  Other Names: Saccharose
  Arms: Sucrose
Dietary Supplement: Sucralose — Subject specific dose of sucralose dissolved in 300 mL tap water.
  Other Names: E955-Sucralose
  Arms: Sucralose

SUMMARY:
The aim of this project is to investigate the reward responses to oral erythritol compared to sucrose and sucralose using flavor preference learning in healthy participants. In addition, the release of GI hormones, glycemic control, appetite-related sensations, and emotional state in response to erythritol will be investigated.

DETAILED DESCRIPTION:
This trial is a randomized, double-blind, cross-over study; the project set-up will be single-centre, national. The study is composed of six visits: one screening visit, one pre-test visit, three conditioning visits, and one post-test visit. The screening and pre-test will last about two hours, the conditioning days and the post-test day about 4 hours each. During the screening participants take part in a 6-n-propylthiouracil (PROP) sensitivity test to exclude potential supertasters. Moreover, the participants will rate explicit liking and explicit wanting of 10 non-caloric flavored and colored beverages in a randomized order (flavor preference learning). The pre-test visit consists of two parts. First, a chemosensory sweetness matching will be performed, during which we will establish dose-response relationships for perceived sweetness of sucrose, erythritol, and sucralose using equisweet watery solutions across a range of concentrations. Second, the participants will perform a triangle test to ensure that they cannot distinguish the matched erythritol and sucralose solutions from a 10% sucrose solution.

During the 3 conditioning visits, participants will be presented with three conditioning trials (at t = 0, 45, and 90min), each consisting of drinking 100mL of the flavored drink (CS) paired with one of the sweet substances (US = erythritol, sucrose, or sucralose).

In post-test visit, preference for each of the 3 flavored CS drinks will be assessed and a computerized forced choice task will be completed by the participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy normal weight participants with a body-mass index (BMI) of 19.0-24.9 kg/m2
* Age 18-55 years
* Stable body weight (±5%) for at least three months
* Able to give informed consent as documented by signature
* 3 drinks rated as neutral and novel (from the flavor preference learning)

Exclusion Criteria:

* Non-taster (deficits of taste and smell) or supertaster
* Fructose intolerance
* Shift worker
* Pre-existing regular consumption of erythritol and/or sucralose and/or aspartame (>1/week)
* Substance abuse (more than 1 glass wine/beer per day; consumption of cannabis, cocaine, heroin, etc.)
* Regular intake of medications, except contraceptives
* Chronic or clinically relevant acute infections
* Pregnancy: although no contraindication, pregnancy might influence metabolic state.
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Pre-existing diet (vegetarian, vegan, sugar free)
* Inability to follow procedures due to psychological disorders or insufficient knowledge of project language (German)
* Calculated dose of erythritol outside the range of 30-60g (per 300mL) (from the sweetness matching)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
Assessment of the change of explicit wanting (reward response) to oral erythritol versus sucrose and sucralose as change from baseline to post-test visit. | from baseline to post-test visit (at t = 0min, t = 45min and t = 90min)
  Beverages are consumed during the screening visit, conditioning visits and the post-test visit. The beverages will be consumed at t = 0min, t = 45min and t = 90min and afterwards explicit wanting will be assessed.
  Explicit wanting of the consumed beverages is assessed by Visual Analogue Scale (VAS) as "How much do you want to drink of the drink". The Visual Analogue Scale consists of a horizontal, unstructured, 10 cm line representing the minimum (0.0 points) labeled with "not much at all" to the maximum rating (10.0 points) labeled with "very much". Participants are instructed to draw a dash in the answer line to indicate the magnitude of their subjective sensation at the present time point.

SECONDARY OUTCOMES:
Effects on reward response - explicit liking | The beverages will be consumed at t = 0min, t = 45min and t = 90min and afterwards explicit liking will be rated.
  Beverages are consumed at the screening visit (during the flavor preference learning), conditioning visits and the post-test visit.
  Explicit liking of the consumed beverages during the screening visit, the conditioning visits and post-test visit is rated from -100 to 100 using the Global Hedonic Intensity Scale (GHIS). The Global Hedonic Intensity Scale ranges from -100 "the most intensive disliking ever experienced" to 100 "most intensive liking ever experienced" and has no anchors and in the middle is 0 as a neutral point. Participants are instructed to draw a dash in the answer line to indicate the magnitude of their subjective liking at the present time point.
Effects on reward response - desire to drink | The beverages will be consumed at t = 0min, t = 45min and t = 90min and afterwards desire to drink will be rated.
  Beverages are consumed at the screening visit (during the flavor preference learning), conditioning visits and the post-test visit.
  During the post-test visit, the desire to drink will be recorded with a 10 cm Visual Analogue Scale (VAS) as "How strong is your desire to drink, that is, to taste and swallow, the rest of the drink RIGHT NOW? (Take a sip of the drink first)". The Visual Analogue Scale consists of a horizontal, unstructured, 10 cm line representing the minimum (0.0 points) labeled with "not strong at all" to the maximum rating (10.0 points) labeled with "very strong". Participants are instructed to draw a dash in the answer line to indicate the magnitude of their subjective sensation at the present time point.
Effects on reward response - implicit wanting | The computerized forced choice task will be performed at t = 135 min during the post-test visit.
  Implicit wanting will be measured at the end of the post-test visit by using a computerized forced choice task. Participants will be shown a paired presentation of three drinks where they have to select their most wanted drink ("select the drink which you would most want to drink right now"). In the four presentation parts, participants will have to choose between e.g. red bull drink vs. diet coke vs. fanta, or between diet coke vs. orange juice vs. ice tea. During the fifth presentation, pictures of the previous conditioned drinks will be shown and participants have to choose the drink which they would most want to drink right now. During the choice task, the chosen drink and the reaction time with which this drink was chosen (implicit wanting) will be measured.
Effects on GI hormone response - GLP-1 | Blood will be drawn at baseline (at t = -1min) and at t = 15, 30, 44, 60, 75, 89, 105, 120, and 134min.
  Plasma GLP-1 will be quantified using a non-radioactive high sensitive sandwich ELISA (Millipore - # EZGLPHS-35K) in the presence of a chemiluminescent substrate.
Effects on GI hormone response - PYY | Blood will be drawn at baseline (at t = -1min) and at t = 15, 30, 44, 60, 75, 89, 105, 120, and 134min.
  PYY-3-36 will be quantified using a non-radioactive high sensitive sandwich ELISA (Millipore - # EZHPYYT66K).
Effects on GI hormone response - CCK | Blood will be drawn at baseline (at t = -1min) and at t = 15, 30, 44, 60, 75, 89, 105, 120, and 134min.
  Plasma cholecystokinin (CCK) levels will be measured with a sensitive radioimmunoassay using a highly specific antiserum (No. 92128)
Effects on GI hormone response - ghrelin | Blood will be drawn at baseline (at t = -1min) and at t = 15, 30, 44, 60, 75, 89, 105, 120, and 134min.
  Octanoylated ghrelin will be measured by a radioimmunoassay with 125I [Tyr24] human ghrelin [1-23] as tracer and a rabbit antibody against human ghrelin [1-8] (final dilution 1/100000), which does not cross-react with desoctanoylated ghrelin.
Effects on glycemic control - plasma glucose | Blood will be drawn at baseline (at t = -1min) and at t = 15, 30, 44, 60, 75, 89, 105, 120, and 134min.
  Glucose will be measured by a glucose oxidase method (Rothen Medizinische Laboratorien AG, Basel, Switzerland).
Effects on glycemic control - plasma insulin | Blood will be drawn at baseline (at t = -1min) and at t = 15, 30, 44, 60, 75, 89, 105, 120, and 134min.
  Insulin will be quantified using a chemiluminescent microparticle immunoassay (chemiflex) reagent kit (#8k41; Abbott) and the relative light units detected by the ARCHITECT optical system (model: CI4100; Abbott).
Effects on glycemic control - plasma c-peptide | Blood will be drawn at baseline (at t = -1min) and at t = 15, 30, 44, 60, 75, 89, 105, 120, and 134min.
  C-peptide will be measured with a commercially available sandwich ELISA kit from Millipore (Millipore - # EZHCP-20K).
Effects on glycemic control - plasma glucagon | Blood will be drawn at baseline (at t = -1min) and at t = 15, 30, 44, 60, 75, 89, 105, 120, and 134min.
  Glucagon concentrations in plasma will be measured after extraction of plasma with 70% ethanol (vol/vol, final concentration). The antibody is directed against the C-terminus of the glucagon molecule (antibody code no. 4305) and therefore mainly measures glucagon of pancreatic origin.
Effects on appetite-related sensations (hunger, thirst, satiety) | Appetite-related sensations will be assessed at t = -1, 0, 15, 30, 44, 45, 60, 75, 89, 90, 105, 120, 134min.
  Hunger, thirst, and satiety are assessed by VASs. VASs consist of a horizontal, unstructured, 10cm line representing the minimum (0.0 points) to the maximum rating (10.0 points). Participants are instructed to draw a dash in the answer line to indicate the magnitude of their subjective sensation at the present time point. The measurement is quantified by the distance from the left end of the line (minimum rating) to the participant's vertical mark.
Emotional state | The emotional state will be assessed at t = -1, 0, 45, 90 min.
  Emotional state will be recorded with the self-assessment manikin (SAM). The self-assessment manikin is a non-verbal pictorial assessment technique using figures that directly measure the pleasure associated with a person's affective reaction to a variety of stimuli. The SAM represent a 9-point scale. The five figures used in this study range from unhappy (0) to happy (9). To indicate their emotional state at a certain time point, participants can select any of the figures or between any of the figures.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Christin Meyer-Gerspach, PD, PhD, Principal Investigator — St. Clara Research Ltd.
Locations (1):
- St. Claraspital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No